CLINICAL TRIAL: NCT03382431
Title: A Single-blind, Placebo Controlled, Randomised Study to Evaluate Antiviral Activity and Safety and Pharmacokinetics of Inhaled PC786 Against Respiratory Syncytial Virus (RSV) in Healthy Adult Subjects in a Virus Challenge Model
Brief Title: A Study of PC786 to Evaluate the Antiviral Activity, Safety and Pharmacokinetics of Multiple Doses in an RSV Challenge Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC_RSV_003; 2017-002563-18 (EudraCT Number)
Record Dates: First submitted 2017-12-08; First posted 2017-12-22 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — PC-786

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC786 (Experimental): Repeat dose
  Interventions: Drug: PC786
- Placebo/vehicle (Placebo Comparator): Repeat dose
  Interventions: Drug: Placebo/vehicle

INTERVENTIONS:
Drug: PC786 — Repeat doses
  Arms: PC786
Drug: Placebo/vehicle — Repeat doses
  Arms: Placebo/vehicle

SUMMARY:
PC786 is a new medicine being developed for treatment of respiratory syncytial virus. The main purpose of this study is to evaluate the antiviral activity of PC786 in healthy adults infected with RSV virus in a viral challenge study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health as determined by the Investigator based on medical history, physical examination, and routine laboratory tests at a screening evaluation.
* Male or female, aged between 18 and 55 years inclusive
* Body weight ≥ 50 kg and Body Mass Index (BMI) ≥ 18 kg/m2 and ≤ 30kg/m2
* Subject must provide written informed consent
* Serosuitable to the challenge virus.

Exclusion Criteria:

* History or evidence of any clinically significant or currently active major clinical illness.
* Any significant abnormality altering the anatomy of the nose or nasopharynx
* Any nasal or sinus surgery within six months of the study
* Abnormal lung function
* Positive human immunodeficiency virus (HIV), active hepatitis A (HAV), B (HBV), or C (HCV) test.
* Presence of cold like symptoms and/or fever on admission for the study
* History or currently active symptoms suggestive of upper or lower respiratory tract infection within 6 weeks of the study
* History of anaphylaxis-and/or a history of severe allergic reaction or significant intolerance to any food or drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
RSV viral load | Baseline to Day 28
  AUC 0-t for RSV viral load measured in nasal washes by reverse transcription quantitative polymerase chain reaction (RT-qPCR)

SECONDARY OUTCOMES:
Number of participants reporting one or more treatment-emergent adverse event (TEAE) | Screening to Day 28
Number of participants who discontinue due to an adverse event | Screening to Day 28
Number of participants who meet the markedly abnormal criteria for 12-lead ECG assessment at least once post dose | Screening to Day 28
Number of participants who meet the markedly abnormal criteria for vital signs assessments at least once post dose | Screening to Day 28
Number of participants who meet the markedly abnormal criteria for safety laboratory assessments at least once post dose | Screening to Day 28
Number of participants who meet the markedly abnormal criteria for spirometry (FEV1 & FVC measured together) assessments at least once post dose | Screening to Day 28
Area under the plasma concentration versus time curve (AUC) of PC786 measured in plasma | Pre-dose and at multiple time points to Day 12
Maximum observed concentration (Cmax) of PC786 measured in plasma | Pre-dose and at multiple time points to Day 12
Time maximum concentration observed (Tmax) of PC786 measured in plasma | Pre-dose and at multiple time points to Day 12
Apparent terminal half life (T1/2) of PC786 measured in plasma | Pre-dose and at multiple time points to Day 12
Determination of nasal concentrations of PC786 | Pre-dose and at multiple time points to Day 28
  PC786 concentrations in mucosal lining fluid collected using synthetic absorptive matrix
Comparison of mucus production following treatment with PC786 or placebo post viral inoculation | Baseline to Day 12
  Reduction in weight of mucus produced post viral infection
Comparison of the effect of treatment with PC786 or placebo on RSV symptoms | Baseline to Day 12
  Composite score of self-reported symptoms on a symptom diary card. Nasal symptoms, sneezing, sore throat, cough, headache, wheezing, chest tightness, shortness of breath, joint aches, feverishness, malaise, earache are assessed using a score of 0 (no symptoms), 1 (just noticeable), 2 (bothersome but able to participate in activities), 3 (bothersome and not able to participate in activities)
Change in viral load measured in nasal wash | Baseline to Day 12
  Change in viral load before first dose of PC786 to Day 12
Time to non-detectability of virus measured in nasal wash | Baseline to Day 12
Peak viral load measured in nasal wash | Baseline to Day 12
Time peak viral load observed measured in nasal wash | Baseline to Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Bryan J Murray, MBBS, Principal Investigator — hVIVO Services Ltd
Locations (1):
- hVIVO Services Ltd, London, United Kingdom

REFERENCES:
- [Derived] DeVincenzo J, Cass L, Murray A, Woodward K, Meals E, Coates M, Daly L, Wheeler V, Mori J, Brindley C, Davis A, McCurdy M, Ito K, Murray B, Strong P, Rapeport G. Safety and Antiviral Effects of Nebulized PC786 in a Respiratory Syncytial Virus Challenge Study. J Infect Dis. 2022 Jun 15;225(12):2087-2096. doi: 10.1093/infdis/jiaa716. PMID 33216113